CLINICAL TRIAL: NCT05421338
Title: A Phase I, Open-label, Single-dose, Single-arm Trial to Investigate Metabolism and Pharmacokinetics of BI 456906 (C-14) Administered Subcutaneously to (Otherwise) Healthy Male Volunteers With Normal Body Weight, Overweight or Obesity
Brief Title: A Study in Healthy Men to Test How BI 456906 is Processed in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0012; 2021-006690-28 (EudraCT Number)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — BI 456906; Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 456906 (C-14) (Experimental)
  Interventions: Drug: BI 456906 (C-14)

INTERVENTIONS:
Drug: BI 456906 (C-14) — BI 456906 (C-14)

SUMMARY:
This trial is intended to examine the basic pharmacokinetics of BI 456906 and total [14C]-radioactivity, including mass balance, excretion pathways and metabolism following a single subcutaneous (SC) dose of BI 456906 (C-14) in (otherwise) healthy male volunteers with normal body weight, overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects with normal Body mass index (BMI) or otherwise healthy male subjects with overweight/obesity according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* BMI of 23.0 to 34.9 kg/m2 (inclusive); body weight of at least 70 kg.
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 45 to 90 mmHg, or pulse rate outside the range of 40 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Fraction of [14C]-radioactivity excreted in urine expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (fe_urine, 0-tz) | up to 7 weeks
Fraction of [14C]-radioactivity excreted in faeces expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (fe_faeces, 0-tz) | up to 7 weeks

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte (Cmax) | up to 22 days
Area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point (AUC0-tz) | up to 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com